CLINICAL TRIAL: NCT01527617
Title: The Effect of Chronic Consumption of a Cranberry Beverage on Inflammation and Oxidative Stress in Healthy But Overweight/Obese Subjects: A Randomized Clinical Trial
Brief Title: Effect of Chronic Consumption of a Cranberry Beverage on Inflammation and Oxidative Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Washington State University (Other); Ocean Spray, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB10178
Record Dates: First submitted 2012-01-30; First posted 2012-02-07 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-06

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Cranberry beverage (Active Comparator)
  Interventions: Other: Cranberry
- Non-cranberry beverage (Placebo Comparator)
  Interventions: Other: Non-Cranberry beverage

INTERVENTIONS:
Other: Cranberry — beverage containing cranberry at a dose of 15.2 ounces per day for 56 days.
  Arms: Cranberry beverage
Other: Non-Cranberry beverage — Placebo Comparator - beverage absent cranberry at a dose of 15.2 ounces per day for 56 days.
  Arms: Non-cranberry beverage

SUMMARY:
The objective of this randomized, double-blind, placebo-controlled, parallel-design clinical trial is to investigate the potential antioxidant benefits of a cranberry beverage. The investigators hypothesize the chronic consumption of this beverage will improve indices of oxidative stress, inflammation, endothelial function, and glucoregulation. The investigators also hypothesize that these benefits will be particularly evident following an oral glucose tolerance test.

ELIGIBILITY:
Inclusion Criteria:

* Men & women, aged 30-70 years
* BMI 27-34.9 kg/m2
* waist:hip ratio > 0.8 for women and > 0.9 for men

Exclusion Criteria:

* Cigarette smoking and/or nicotine replacement use within last 6 months
* Individuals taking estrogen or testosterone
* Use of cholesterol-lowering medications
* Use of blood pressure-lowering medications
* Regular use (> 1x/wk) of any stomach acid-lowering medications or laxatives (including fiber supplements)
* Cardiovascular (heart) disease
* Gastrointestinal disease
* Kidney disease
* Endocrine disease: including diabetes, untreated thyroid disease
* Rheumatoid arthritis
* Immune deficiency conditions
* Active treatment for any type of cancer, except basal cell carcinoma, within 1 year prior to study admission
* Systolic blood pressure > 139 mmHg and/or diastolic blood pressure > 89 mmHg
* Regular use of systemic steroids, oral or injectable
* Regular daily intake of ≥ 2 alcoholic drinks
* Infrequent (< 3/week) or excessive (> 3/d) number of regular bowel movements
* Gain or loss of ≥ 5% of body weight in the last 6 months
* Pregnancy
* Strict vegetarians
* No dietary supplements, including those containing any vitamins, minerals, herbs, plant concentrates (including garlic, gingko, St. John's wort) homeopathic remedies, probiotics, or fish oil (including cod liver oil), for one month prior to study admission

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2012-02; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Change in biomarkers of inflammation compared with placebo | Baseline and 8 weeks
Change in biomarkers of oxidative stress compared with placebo. | Baseline and 8 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts
  - Washington State University, Pullman, Washington